CLINICAL TRIAL: NCT04453995
Title: A Follow-up of the Influencing Factors of Dyskinesia in Patients With Parkinson's Disease
Acronym: PDDIFFU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Second Affiliated Hospital of Soochow University (Other); The Affiliated BenQ Hospital of Nanjing Medical University (Unknown); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Zhejiang Provincial Tongde Hospital (Other); Shaoxing Hospital of Traditional Chinese medicine (Unknown); The First People Hospital of Hangzhou Lin An District (Unknown)
Responsible Party: Sponsor
Other Study IDs: XH-19-014
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease; Dyskinesias
Keywords: Parkinson disease; Dyskinesia; follow up
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — every participant would be request for provide 2 ml blood for extracting the DNA sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson' patients who have not had dyskinesia would be observed for 2 years in a multicenter prospective study with the purposes to clarify the predicting factors of dyskinesia.

DETAILED DESCRIPTION:
Parkinson' patients with daily levodopa dosage above 200mg and no dyskinesia would be recruited into the study. They would be observed for two years for analyzed the predicting factors of dyskinesia. At the baseline, demographic information, Clinical information, blood sample, picture of tongure coating would be collected at the baseline. All participants were evaluated every three months for two years. The severity of motor symptoms were evaluated every 6 months.

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients have been clinically diagnosed with Parkinson disease at the recruitment.

2) Patients have received Levodopa treatment with the daily dosage above 200mg.

Exclusion Criteria:

* 1) be suspicious of atypical Parkinson or other Parkinson syndrome. 2) have experienced dyskinesia. 3) incorporation to the investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: a 2 years prospective study to identify the predicting factors of dyskinesia in Parkinson' patients that have received Levodopa treatment.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
the occurrence of dyskinesia and its related predicting factors | The data would be analyzed within 9 months of the study completion. The outcome would be reported within 1 year of the the study completion.
  to evaluate the occurrence of dyskinesia during the 2 years of follow-up and identify its predicting factors of dyskinesia

SECONDARY OUTCOMES:
to evaluate patients ' living quality and the severity of non motor symptoms during the 2 years of follow-up | The data would be analyzed within 9 months of the study completion. The outcome would be reported within 1 year of the the study completion.
  to evaluate patients ' living quality and the severity of non motor symptoms during the 2 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: zhenguo Liu, Ph.D., Study Chair — Xinhua hosipital affiliated to Shanghai Jiaotong university school of medicine
Locations (1):
- Xinhua hospital affiliated to Shanghai jiaotong university school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
There would be digital data of all the information that collected in the study. But it is still unknown that the data would be available freely